CLINICAL TRIAL: NCT00398255
Title: Internet Arthritis Self-Management Study
Brief Title: Healthier Living With Arthritis Online Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NIH-AR43538
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Fibromyalgia
Keywords: arthritis; self management; patient education
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Fibromyalgia; Arthritis | interventions — Self-Management

INTERVENTIONS:
Behavioral: self-management program

SUMMARY:
Individuals with with arthritic conditions (rheumatoid arthritis, osteoarthritis, or fibromyalgia) and internet and email access were randomized to receive an internet-based arthritis self-management program (treatment group) or to continue with usual care (control group). Questionnaires measuring health indicators, health behaviors, self efficacy and health care utilization were administered at baseline, six months and one year after the course. It was hypothesized that those participating in the course would have better outcomes than the control group at six months and one year.

DETAILED DESCRIPTION:
An internet-based arthritis self-management program was developed based on the widely used small-group arthritis self-management program. Individuals with arthritis were recruited via established websites, on-line newsletters, discussion groups, calendar announcements and articles in newspapers, and asked to go to the project website. Subjects who filled out an informed consent and met all of the following criteria were invited to enroll:

1. At least 18 years of age
2. A physician's diagnosis of osteoarthritis, rheumatoid arthritis or fibromyalgia.
3. Not have been in active treatment for cancer for one year.
4. Not participated in the small group Arthritis Self-Management or Chronic Disease Self-Management Program

Those eligible and wishing to continue were randomized to receive the internet-based arthritis self-management program (treatment group) or to continue with usual care (control group). On-line questionnaires were administered at baseline, six months and twelve months after the program. Measures included health indicators, health behaviors, self efficacy and health care utilization. It is hypothesized that course participants, compared to the usual-care control group, will show statistically significant improvements (using Analyses of Covariance and Logistic Regressions) in outcome variables and that the improvements will be associated with increased self-efficacy for management of arthritis.

ELIGIBILITY:
Inclusion Criteria:

* arthritic condition (osteoarthritis, rheumatoid arthritis or fibromyalgia)
* internet access and ability to use computer

Exclusion Criteria:

* active treatment for cancer
* taken small group arthritis self-management program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Health Distress Scale at six months and one year
Activities Limitation Scale at six months and one year
Self Efficacy for Management of Arthritis Scale at six months and one year
Stretching and strengthening exercise at six months and one year
Visits of Physicians at six months and one year

SECONDARY OUTCOMES:
Self-Reported General Health at six months and one year
Visual Numeric Pain at six months and one year
Visual Numeric Fatigue at six months and one year
Disability at six months and one year
Aerobic Exercise at six months and one year
Communication with Physician at six months and one year
Cognitive Sympton Management at six months and one year
Emergency Department Visits at six months and one year
Nights in Hospital at six months and one year

CONTACTS AND LOCATIONS:
Overall Officials: Kate R. Lorig, DrPh, Principal Investigator — Stanford School of Medicine
Locations (1):
- Stanford University School of Medicine Patient Education Center, Palo Alto, California, United States

REFERENCES:
- [Derived] Lorig KR, Ritter PL, Laurent DD, Plant K. The internet-based arthritis self-management program: a one-year randomized trial for patients with arthritis or fibromyalgia. Arthritis Rheum. 2008 Jul 15;59(7):1009-17. doi: 10.1002/art.23817. PMID 18576310